CLINICAL TRIAL: NCT06939790
Title: Digital Cognitive-behavioral Therapy for Insomnia: a Randomized Controlled Trial to Improve Cost-effectiveness and Treatment Outcomes
Brief Title: Digital Cognitive-behavioral Therapy for Insomnia: a Randomized Controlled Trial
Acronym: DCBT-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Ferini Strambi, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CET 129-2025; CET 129-2025 (Other: CET Lombardia 1)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Insomnia
Keywords: Sleep; Insomnia; Cognitive-Behavioral Therapy for Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Cognitive-Behavioral Therapy for Insomnia (dCBT-I) (Experimental): The digital CBT-I (dCBT-I) is a self-guided online program replicating the structure and content of standard face-to-face CBT-I, aiming to offer a more accessible treatment for chronic insomnia. It includes video lessons, interactive exercises, and relaxation techniques, with core components such as sleep education, sleep restriction, stimulus control and cognitive restructuring. Supervision is provided through periodic check-ins.
  Interventions: Behavioral: Digital Cognitive-Behavioral Therapy for Insomnia (dCBT-I)
- standard face-to-face group-based Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): The control group will receive standard face-to-face group-based CBT-I, the current gold-standard treatment for chronic insomnia. Delivered by trained professionals, the intervention includes seven structured sessions covering core components such as sleep education, sleep restriction, stimulus control cognitive restructuring, and relaxation techniques. Sessions last about 90 minutes and aim to improve sleep quality through evidence-based strategies.
  Interventions: Behavioral: standard face-to-face group-based Cognitive-Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Digital Cognitive-Behavioral Therapy for Insomnia (dCBT-I) — The digital CBT-I (dCBT-I) is a self-guided online program replicating the structure and content of standard face-to-face CBT-I, aiming to offer a more accessible treatment for chronic insomnia. It includes video lessons, interactive exercises, and relaxation techniques, with core components such as sleep education, sleep restriction, stimulus control and cognitive restructuring. Supervision is provided through periodic check-ins.
  Arms: Digital Cognitive-Behavioral Therapy for Insomnia (dCBT-I)
Behavioral: standard face-to-face group-based Cognitive-Behavioral Therapy for Insomnia (CBT-I) — The control group will receive standard face-to-face group-based CBT-I, the current gold-standard treatment for chronic insomnia. Delivered by trained professionals, the intervention includes seven structured sessions covering core components such as sleep education, sleep restriction, stimulus control, cognitive restructuring, and relaxation techniques. Sessions last about 90 minutes and aim to improve sleep quality through evidence-based strategies.
  Arms: standard face-to-face group-based Cognitive-Behavioral Therapy for Insomnia (CBT-I)

SUMMARY:
The study investigates whether online Cognitive-Behavioral Therapy for insomnia is as effective as the standard in-person group treatment, using clinical and sleep-related outcomes in adult patients.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) in Italian, comparing it to the traditional face-to-face group-based CBT-I. Sixty adults with chronic insomnia will be randomized to one of the two interventions, with assessments conducted pre- and post-treatment through validated questionnaires and objective sleep monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic insomnia Individuals aged 18 to 75 years Signed informed consent form (ICF) prior to study participation

Exclusion Criteria:

* Diagnosis of comorbid sleep disorder (e.g. obstructive sleep apnea) Diagnosis of mental disorder in comorbidity Physical problems that may alter and dysregulate sleep Pregnancy and breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess whether the benefits of dCBT-I are comparable with CBT-I treatment in standard group mode | Change from baseline to post-treatment (2 months)
  Comparison at Insomnia Severity Index (ISI) questionnaire between the two groups evaluated at baseline and post-treatment.

IPD SHARING:
Plan to Share IPD: No